CLINICAL TRIAL: NCT00236327
Title: Evaluation of the Efficacy and Safety of Transdermal Fentanyl in Patients Suffering From Chronic Cancer Pain in an Ambulatory Setting
Brief Title: Evaluation of the Efficacy and Safety of Fentanyl Delivered by Adhesive Skin Patch in Out-Patients With Chronic Cancer Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor discontinued the study following the discovery of a number of incompletely sealed batches that were unusable.
Sponsor: Janssen Cilag S.A.S. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002920
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Pain
Keywords: Fentanyl; Analgesia; Pain; Cancer pain; Opioid analgesia; Transdermal fentanyl; Patient-controlled analgesia
MeSH Terms: conditions — Pain; Agnosia; Cancer Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fentanyl

SUMMARY:
The purpose of this study is to determine the safety and efficacy of pain control by fentanyl, administered via adhesive skin patches, at doses of 25 to 100 micrograms per hour in 80 out-patients with intense chronic cancer pain. Higher doses are allowed by permission of the investigator and rescue oral morphine medication is allowed.

DETAILED DESCRIPTION:
Patients with cancer pain are frequently under-medicated with morphine. This is a 56-day open-label study of the efficacy and safety of self-administered fentanyl skin patches for cancer pain control in patients in the home-care setting not previously using morphine. The first 15 days of the study are for dose stabilization and the rest of the study assesses pain control and quality of life at stable doses of medication. The dose is determined by the patient with oversight by the investigator, and rescue oral morphine medication can be used when necessary. The patient records all medication use in a diary and fills out questionnaires concerning pain control, intestinal function (constipation) and overall quality of life. The hypothesis is that patients will be able to control their cancer pain by self-administering transdermal fentanyl at home and that they will well tolerate the medication.

Individualized doses, with a target dose of 25 to 100 micrograms per hour of fentanyl for 56 days via skin patches applied every 3 days to deliver 25 to 100 micrograms of fentanyl per hour per patch; oral morphine as rescue medication for pain.

ELIGIBILITY:
Inclusion Criteria:

* Less than a month of opioid treatment over the past 3 months
* Proven cancer and chronic stable, cancer-related pain
* Pain control medication (aside from opioids) at the maximum authorized dose in the 24-hours preceding the first study visit
* A pain score of at least 4 on the VAS scale and pain that justifies intervention by opium-derived drugs in the opinion of the investigator

Exclusion Criteria:

* Liver or kidney problems
* Previous heart, lung or nervous disorders
* Allergy to fentanyl
* Skin condition that might interfere with absorption of the fentanyl through the skin
* Surgery or chemotherapy in the month preceding the study or scheduled during the 56 days of the study
* History of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-06; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Pain control level using a visual analog scale (VAS) at various time points and at the end of 56-day study. Percent pain reduction and percentage of patients having a score of 4 or lower compared to the baseline. Use of rescue medication.

SECONDARY OUTCOMES:
Constipation and recorded use of laxatives, patient-assessed quality of life obtained by questionnaires and overall tolerance assessed at the end of 56-day study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A.S. Clinical Trial, Study Director — Janssen Cilag S.A.S.

REFERENCES:
- See also: Assessment of the efficacy and tolerance of transdermal fentanyl in patients with chronic cancer pain in outpatient medicine — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=272&filename=CR002920_CSR.pdf